CLINICAL TRIAL: NCT04204135
Title: The Course of Hip Flexion Weakness Following LLIF or ALIF
Status: Enrolling by invitation | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16081205
Record Dates: First submitted 2019-08-20; First posted 2019-12-18 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Degenerative Disc Disease; Herniated Nucleus Pulposus; Spondylolisthesis
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: LLIF or ALIF procedures — LLIF or ALIF procedures

SUMMARY:
The purpose of this study is to assess the course of hip weakness after LLIF or ALIF procedures. These outcomes include measures of hip strength using a dynamometer, which is a device used to measure muscle strength. While it is known that people experience temporary hip and leg weakness after an LLIF or ALIF, the exact timing of when hip and leg strength is regained after an LLIF or ALIF is not known.

ELIGIBILITY:
Inclusion Criteria:

* 1-, 2-, or 3-level L2L3, L3L4, or L4L5 LLIF or ALIF for degenerative pathology including radiculopathy, neurogenic claudication, intervertebral disc disease, facet joint disease, degenerative spondylolisthesis, degenerative myelopathy degenerative kyphosis, and scoliosis
* Back and/or leg pain
* Failed at least 6 months of conservative treatment

Exclusion Criteria:

* Older than 65 years of age
* Prior spinal fusion surgery
* Greater than Grade 2 spondylolisthesis
* Greater than 10° scoliosis
* History of spinal infection

Max Age: 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing LLIF or ALIF procedures
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2018-10-04 (Actual); Primary Completion 2027-09-04 (Estimated); Study Completion 2027-11-04 (Estimated)

PRIMARY OUTCOMES:
Hip flexion and knee extension strength as measured by the Lafayette Instrument Manual Muscle Testing Device (Dynamometer). | Assessing changes in hip flexion and leg extension strength from the preoperative baseline to postoperative measurements taken at 6 weeks, 12 weeks and 6 months following lumbar fusions.
  Using a Lafayette Instrument Manual Muscle Testing Device (Dynamometer), we will be measuring the force in pounds a given patient can exert upon hip flexion and knee extension at the preoperative timepoint and 6 weeks, 12 weeks and 6 months postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No